CLINICAL TRIAL: NCT07338279
Title: Parvovirus B19 Infection in Pregnancy: Clinical Manifestations and Fetus/Newborn Outcome
Acronym: ParvoPre
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); ASST Fatebenefratelli Sacco (Other); Fondazione IRCCS San Gerardo dei Tintori (Other); Asst Degli Spedali Civili Di Brescia (Other)
Responsible Party: Principal Investigator, Daniele Lilleri, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: ParvoPre
Record Dates: First submitted 2025-11-19; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Parvovirus B19 Infection; Pregnancy
MeSH Terms: conditions — Erythema Infectiosum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

INTERVENTIONS:
Other: Collection of clinical data. — Observational study

SUMMARY:
The goal of this observational study is to define the rate of intrauterine parvovirus B19 infection and fetal/newborn complications after parvovirus B19 infection of pregnant women. Secondary objectives are risk factors, pregnancy outcomes, long-term sequelae and efficacy of the management interventions.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women >18 years with parvovirus B19 infection and their neonates.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of fetuses/newborns with intrauterine B19V infection. | From diagnosis of parvovirus B19 infection in pregnancy to 24/48 hours of life of the newborn.
Percentage of fetuses/newborns with complications due to B19V intrauterine infection. | From diagnosis of parvovirus B19 infection in pregnancy to 24/48 hours of life of the newborn.

SECONDARY OUTCOMES:
Percentage of women with symptomatic B19V infection. | At diagnosis of parvovirus B19 infection in pregnancy
Percentage of fetuses with B19V disease. | From diagnosis of parvovirus B19 infection in pregnancy to delivery.
  The following findings will be considered: anemia, hydrops, ascites, pericardial effusion, pleural effusion, subcutaneus oedema, cardiomegaly, placental thickening, cerebral abnormalities, growth retardation.
Percentage of fetuses receiving intrauterine transfusion. | From diagnosis of parvovirus B19 infection in pregnancy to delivery.
Percentage of newborns with B19V disease. | From diagnosis of parvovirus B19 infection in pregnancy to 20/30 days of life of the newborn.
  The following signs/symptoms will be considered: anemia, paleness, petechiae, purpura, icterus, hepato-splenomegaly, ascites, hydrops, pleural effusion, pericardial effusion, neurologic abnormalities.
Percentage of infants with neurologic abnormalities. | From birth to 2 years of life.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - ASST degli Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza

IPD SHARING:
Plan to Share IPD: Undecided